CLINICAL TRIAL: NCT03908710
Title: A Prospective Trial of Home Blood Pressure Levels in Hypertensive Participants Using the ACCUMBO Telemedicine Device
Brief Title: The Accumbo Home Blood Pressure Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Accumbo AB (Other)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Accumbo AB (Accumbo)
Record Dates: First submitted 2019-04-07; First posted 2019-04-09 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Hypertension,Essential
Keywords: Home blood pressure monitor; Telemedicine; mHealth; eHealth
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- home Home blood pressure levels in hypertensive participants (Other): Only one arm. No control group.
  Interventions: Other: Treatment of hypertension using blood pressure self-measurement at home

INTERVENTIONS:
Other: Treatment of hypertension using blood pressure self-measurement at home — The primary aim of the present study is to investigate whether home blood pressure recording via Bluetooth and continuous communication between doctor and patient will give improved blood pressure values when comparing the initial values with the blood pressure values recorded after 3 months. Secondary examinations include treatment of hypotension and adverse events, the patient's experience, the user's potential problems with the blood pressure cuff, app downloading, problems with history issues or problems with technical

SUMMARY:
Aim of the study was to investigate a new clinical medical system for treatment of hypertension with a clinical decision system,a smartphone patient app and a home blood pressure monitor.

DETAILED DESCRIPTION:
Despite the extensive knowledge of the importance of treating and thus preventing complications of hypertension, the incidence of high blood pressure is increasing, and it is still the main cause of cardiovascular disease and premature death, partly due to deficiencies in preventive care and control of the disease in an aging world. Blood pressure values obtained by self-measurement at home (HBPM) have been shown to predict the cardiovascular prognosis equally well as or better than blood pressure values obtained in the clinic (CBPM) in several observational studies. Aim of the present study was to investigate a new clinical medical system for treatment of hypertension with a clinical decision system and a electronic health record, a patient app and a home blood pressure monitor. " The patient app and the doctor's record reflect each other and basically contain the same information. Doctors can treat their patients remotely and the patients are able to manage some health issues by themselves by using the applications. Some patients need the physical examination. We therefore included patients after a so-called triage step with medical questions.

ELIGIBILITY:
Inclusion Criteria:

* Primary hypertension
* Smartphone at home

Exclusion Criteria:

* Secondary hypertension,
* previous stroke,
* myocardial infarction,
* known heart failure,
* known cardiac arrhytmia,
* known servere renal failure,
* known dementia

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in mean home blood pressure (systolic and diastolic blood pressure mmHg) during the trial using automatic oscillometric blood pressure monitor | 3 months
  We investigate if the blood pressure is better in the end of the study compared with the start
Patient experience | 3 months
  We investigate how the patients experience the medical technology system and the treatment using a questionnaire

SECONDARY OUTCOMES:
Hypotension | 3 months
  We investigate how many patients have hypotension/ortosstatism in the beginning of the study compared in the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Martin Carlsson, MD,PhD, Principal Investigator — Accumbo AB
Locations (1):
- Martin Carlsson,, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.accumbo.se